CLINICAL TRIAL: NCT06796309
Title: Assessment of Rural Health Care: Introduction of the TRAK Digital Tool for Quality and Accessible Medical Care
Brief Title: Assessment of Rural Health Care: Implementing TRAK Digital Tool for Quality and Accessible Services
Acronym: TRAK-RURAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trak Health Solutions S.L. (Industry)
Collaborators: University Hospital Gregorio Marañón (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRAK-RURAL
Record Dates: First submitted 2025-01-07; First posted 2025-01-28 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Shoulder Pain
Keywords: shoulder pain; telerehabilitation; telemedicine; exercise program; physiotherapy; healthcare personnel
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Prospective experimental study with 95 participants (15 from Population 1; 80 from Population 2) included based on compliance with inclusion and exclusion criteria.
  Population 1:
  Fifteen healthcare professionals will be recruited.
  The intervention targets patients with musculoskeletal pathologies using randomized allocation into two groups: a treatment group utilizing Trak and a control group following conventional rehabilitation methods.
  Population 2:
  Eighty patients will be randomly assigned to the experimental or control group in a 1:1 ratio.
Who Masked: Participant
Masking Description: Randomization is achieved through permuted block randomization with a 1:1 allocation ratio, ensuring balance. The intervention includes remote rehabilitation exercises supported by healthcare professionals, with outcomes assessed independently for both populations (healthcare staff and patients).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TRAK treatment group (Population 2) (Experimental): Patients will use Trak platform for 8 weeks (2 months) for their exercise program. The use of the tool involves performing the corresponding therapeutic exercise program through it. The frequency of the exercises will be determined by the healthcare professional responsible for the patient, based on the needs identified during the assessment, ranging from 3 to 7 days per week.
  Interventions: Other: Trak Telerehabilitation Platform
- Control Group (Population 2) (Active Comparator): Patients in the control group will undergo the same rehabilitation period (8 weeks) but following standard clinical practice.
  Interventions: Other: Conventional Rehabilitation Program
- Healthcare professional Group (Population 1) (Other): Healthcare professionals who will have access to the tool to prescribe exercise sessions for their patients, monitor their progress, adapt and modify the exercise program, communicate with patients to address their questions, and track their progress over time.
  Interventions: Other: Trak Telerehabilitation Platform

INTERVENTIONS:
Other: Trak Telerehabilitation Platform — The exercise protocol designed is carried out through TRAK, the digital rehabilitation tool.
  Arms: Healthcare professional Group (Population 1); TRAK treatment group (Population 2)
Other: Conventional Rehabilitation Program — Exercise protocol with the methodology of conventional clinical practice.
  Arms: Control Group (Population 2)

SUMMARY:
This clinical trial aims to analyze the usability and degree of satisfaction of two populations, healthcare personnel (Population 1) in rural areas and their patients (Population 2), with the TRAK tele-rehabilitation tool.

Participants will undergo telerehabilitation treatment through the TRAK platform for eight weeks (treatment group) or follow an at home exercise protocol (control group).

DETAILED DESCRIPTION:
The recruitment process for this study is aimed at patients with shoulder pain (population 2) and healthcare personnel (population 1).

After the initial screening, individuals who meet the study's predefined inclusion criteria will be invited to participate. Before enrollment, written informed consent will be obtained from all participants, ensuring ethical compliance and respect for individual autonomy.

The healthcare personnel (population 1) will use Trak during the entire study period, from the time of entry into the study to the time of exit.

The study cohort will consist of patients randomly assigned to the experimental group (EG) and the control group (CG) on the first in person visit for the population 2 (patients). Regardless of group assignment, all patients will undergo baseline health assessments, ensuring that their individual needs are met. The satisfaction questionnaire will be deferred until post-intervention for both groups.

Participants in both groups will begin by filling out the Quality of Life Scale (EuroQol 5). and Shoulder Functional Assessment Scale (SPADI-Br) on the first visit.

In the case of the treatment group (EG), the participants will use the platform following the treatment prescribed by their health professionals for a period of 2 months. in the case of the control group (CG), the patients will follow the usual clinical practice treatment (they will receive the exercise protocol in paper format).

At the end of the treatment period, a final face-to-face visit will be made.

Patients (population 2) will undergo 8 weeks of treatment through the TRAK tool (https://www.trakphysio.com/es/) in the EG. Patients from the EG will carry out the treatment through the platform at home, and those from the CG will follow an on paper exercise protocol based on the usual (in-person) clinical practice methodology. Both groups will perform exercises in these rehabilitation sessions to improve shoulder mobility.

The results will be evaluated using different métrics, such as Telemedicine Usability Questionnaire (TUQ) and Telemedicine Satisfaction and Usefulness Questionnaire (TSUQ), wich are the main ones, number of patients using the platform, the EuroQol-5D and the shoulder functional evaluation scale (SPADI-Br). These scales will be completed on paper at the beginning and end of the study for both groups.

ELIGIBILITY:
Inclusion Criteria population 1:

* They carry out their activity in a rural environment.
* That they know how to use the tool.
* That they have a device with which to use the tool.
* That they have an e-mail address.
* That they have an Internet connection.
* That they have signed the informed consent form.

Exclusion Criteria population 1:

* N/A

Inclusion Criteria population 2:

* Seniors.
* Patients with omalgia of more than 6 months of evolution.
* Who have a device with which to use the tool.
* Who have a device with which to use the tool.
* Who have an Internet connection.
* Who have an e-mail address.
* Who have signed the informed consent form.

Exclusion Criteria population 2:

* Patients with cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Telemedicine Usability Questionnaire (TUQ). | Last visit, week 8
  The TUQ is a questionnaire specifically designed to measure (from 17 to 109 points) the usability of telemedicine systems from the perspective of healthcare personnel.
Telemedicine Satisfaction and Usefulness Questionnaire (TSUQ). | Last visit, week 8
  Scale designed to evaluate the satisfaction and usefulness perceived by telemedicine users from 17 to 85 points.

SECONDARY OUTCOMES:
European quality of life 5 dimension questionnaire (EuroQol-5D) | week 1 and 8
  Generic and standardized questionnaire developed to describe and assess health-related quality of life. This questionnaire has an EVA scale from 0 to 100 and 5 questions that gives a 5 digit patient profile (From 11111 if the patients does not have problems on any item to 33333 if the patients have severe problems). The items valued are personal care, daily activities, mobility, pain and anxiety/depression.
Focus on Shoulder Pain and Disability Index (SPADI-Br). | week 1 and 8
  The SPADI-Br was designed to evaluate the degree of shoulder pain and discomfort in performing activities of daily living from 0 to 130 points.
Number of patients using the platform | week 8
  The total number of patients who are using the TRAK platform.

CONTACTS AND LOCATIONS:
Overall Officials: ANA VADILLO CORTÁZAR, Principal Investigator — Hospital Universitario del Sureste
Locations (1):
- Hospital Universitario del Sureste, Madrid, Spain